CLINICAL TRIAL: NCT03204903
Title: Laser Acupuncture Therapy in Patients With Dry Eye: A Two-center Randomized Controlled Trial
Brief Title: Laser Acupuncture for Dry Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMRPG8F0551; 201600333A3 (Other: Chang Gung Medical Foundation Institutional Review Board)
Record Dates: First submitted 2017-05-21; First posted 2017-07-02 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Dry Eye
Keywords: Dry eye; Laser acupuncture; Traditional Chinese medicine
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Subjects with dry eye are enrolled at two ophthalmic centers and randomly assigned to a laser acupuncture group and control group under conventional treatment with artificial tears. The subjects are treated at acupoints including BL2, TE23, ST2, LI4, ST36, and GB37 using verum or sham laser acupuncture during 3 sessions per week. After 4 and 12 weeks of treatment, the differences in the Tear film break-up time, Schirmer test, visual analogue scale, Ocular Surface Disease Index of the patients are analyzed, and compared between the laser acupuncture and control groups using paired t-test and one way ANOVA.
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham laser acupuncture: laser acupuncture without laser output.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser acupuncture (Experimental): The subjects are treated at acupoints including BL2, TE23, ST2, LI4, ST36, and GB37 using laser acupuncture during 3 sessions per week for 12 weeks.
  Interventions: Procedure: Laser acupuncture
- Sham laser acupuncture (Sham Comparator): The subjects are treated at acupoints including BL2, TE23, ST2, LI4, ST36, and GB37 using sham laser acupuncture (without laser output) during 3 sessions per week for 12 weeks.
  Interventions: Procedure: Sham laser acupuncture

INTERVENTIONS:
Procedure: Laser acupuncture — Subjects were treated 3 times per week for 12 weeks with the LaserPen (GaAlAs laser diode, 810 nm, 150 mW, pulsed waves), which delivered 0.375 J of energy (5 s) to BL2, TE23, ST2, LI4, ST36, and GB37.
  Arms: Laser acupuncture
Procedure: Sham laser acupuncture — Subjects were treated 3 times per week for 12 weeks with the LaserPen without laser output (5 s) to BL2, TE23, ST2, LI4, ST36, and GB37.
  Arms: Sham laser acupuncture

SUMMARY:
Subjects with dry eye are enrolled at two ophthalmic centers and randomly assigned to a laser acupuncture group and control group under conventional treatment with artificial tears. The effects of laser acupuncture therapy for patients with dry eye are investigated.

DETAILED DESCRIPTION:
Objective: Dry eye is a common ophthalmologic disorder causing ocular discomfort in daily life. The investigators aim to investigate the effects of laser acupuncture therapy for patients with dry eye.

Methods: 200 subjects with dry eye are enrolled at two ophthalmic centers and randomly assigned to a laser acupuncture group and control group under conventional treatment with artificial tears. The subjects are treated at acupoints including BL2, TE23, ST2, LI4, ST36, and GB37 using verum or sham laser acupuncture during 3 sessions per week. After 4 and 12 weeks of treatment, the differences in the Tear film break-up time, Schirmer test, visual analogue scale, Ocular Surface Disease Index of the patients are analyzed, and compared between the laser acupuncture and control groups using paired t-test and one way ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* 20 < age < 65, with aggravated dry eye (one or both eyes), evaluated by ophthalmologist and provides informed consent.
* Tear film break-up time < 10 s
* Schirmer's strips with anesthesia < 5mm/ 5min

Exclusion Criteria:

* presence of eye lesions, received operation for eye during the past three months, combination of other ophthalmic medication, or using contact lens
* pregnancy, diabetes mellitus, vitamin A deficiency, sequelae of Bell's palsy, hemodialysis
* critical illness such as Stevens-Johnson syndrome, etc
* has taken or needs active treatment (including Chinese medicine)
* presence of a pacemaker; history of seizure or epilepsy; using immunosuppressants; cancer; infectious disease of skin
* does not meet the physician's assessment for recruitment
* lack of informed consent.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index | 12 weeks
  The Ocular Surface Disease Index (OSDI) is a 12-item scale for the assessment of symptoms related to dry eye disease and their effect on vision.

SECONDARY OUTCOMES:
Schirmer test | 12 weeks
  A Schirmer's test is used to assess how quickly the eyes produce tears.
Visual analogue scale of eye discomfort | 12 weeks
  A 10-cm visual analog scale (0-10 points, least to greatest discomfort intensity, VAS) was used to measure the intensity of eye discomfort.
Tear film break-up time | 12 weeks
  Tear film break-up time (TFBUT) measures the time required for tears to naturally evaporate and diffuse after blinking.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shin MS, Kim JI, Lee MS, Kim KH, Choi JY, Kang KW, Jung SY, Kim AR, Kim TH. Acupuncture for treating dry eye: a randomized placebo-controlled trial. Acta Ophthalmol. 2010 Dec;88(8):e328-33. doi: 10.1111/j.1755-3768.2010.02027.x. Epub 2010 Nov 10. PMID 21070615
- [Derived] Hu WL, Yu HJ, Pan LY, Wu PC, Pan CC, Kuo CE, Tseng YJ, Hung YC. Laser Acupuncture Improves Tear Film Stability in Patients with Dry Eye Disease: A Two-Center Randomized-Controlled Trial. J Altern Complement Med. 2021 Jul;27(7):579-587. doi: 10.1089/acm.2020.0524. Epub 2021 Apr 27. PMID 33904792
- [Derived] Hu WL, Wu PC, Pan LY, Yu HJ, Pan CC, Hung YC. Effect of laser acupuncture on dry eye: A study protocol for a 2-center randomized controlled trial. Medicine (Baltimore). 2018 Jun;97(22):e10875. doi: 10.1097/MD.0000000000010875. PMID 29851803